CLINICAL TRIAL: NCT04823052
Title: A Phase 2, Placebo-controlled, Adaptive Design Study to Explore the Safety and Efficacy of Sulindac (HLX-0201) and Gaboxadol (HLX-0206) and Possible Other Treatments in Adolescent and Adult Males With Fragile X Syndrome (FXS)
Brief Title: Investigation of Sulindac (HLX-0201) and Gaboxadol (HLX-0206) in Male Fragile X Syndrome Patients Aged 13-40
Acronym: IMPACT-FXS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Healx has experienced delays to the site activation of the study and this has had an adverse impact on the recruitment timeline which is delaying the progress of other projects in our FXS programme.
Sponsor: Healx Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX002-0201
Record Dates: First submitted 2021-03-24; First posted 2021-03-30 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome; FXS
MeSH Terms: conditions — Fragile X Syndrome | interventions — Sulindac; gaboxadol

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to 1 of 4 treatment arms. All treatment arms will be conducted in parallel. Fifteen subjects will be included in each arm. The study treatment will be blinded to patients, carers and physicians.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): One capsule, twice a day
  Interventions: Drug: Placebo
- Sulindac (HLX-0201), dose strength 1 (Active Comparator): One capsule, twice a day
  Interventions: Drug: Sulindac (HLX-0201), dose strength 1
- Sulindac (HLX-0201), dose strength 2 (Active Comparator): One capsule, twice a day
  Interventions: Drug: Sulindac (HLX-0201), dose strength 2
- Gaboxadol (HLX-0206) (Active Comparator): One capsule, twice a day
  Interventions: Drug: Gaboxadol (HLX-0206)

INTERVENTIONS:
Drug: Sulindac (HLX-0201), dose strength 1 — Sulindac (HLX-0201) Capsule
  Arms: Sulindac (HLX-0201), dose strength 1
Drug: Sulindac (HLX-0201), dose strength 2 — Sulindac (HLX-0201) Capsule
  Arms: Sulindac (HLX-0201), dose strength 2
Drug: Placebo — Placebo Capsule
  Arms: Placebo
Drug: Gaboxadol (HLX-0206) — Gaboxadol (HLX-0206) Capsule
  Arms: Gaboxadol (HLX-0206)

SUMMARY:
This study is to investigate the safety, tolerability and efficacy of Sulindac (HLX-0201) and Gaboxadol (HLX-0206) in males with Fragile X Syndrome (FXS) with confirmed full FMR1 mutation treated over a 10 week period in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject consents to participate, or if the subject are not the subjects own legal guardian, offers assent supported by legally authorized representative consent. Caregiver also commits to the study requirements prior to any study-related procedures
* Willing and able to comply with the study procedures as specified in the protocol and to comply with the study drug administration
* Subject and caregiver are both able to understand the spoken national language clearly and caregiver can read and write to complete study assessments
* Males aged 13 to 40 years (inclusive)
* Has FXS with molecular genetic confirmation of the full FMR1 mutation (>200 CGG repeats). May have been confirmed historically or at Screening
* Weight ≥45 kg
* CGI-S score ≥4
* Is in general good health as deemed by the Investigator, determined by physical examination, medical history and laboratory tests
* If receiving sertraline, is on a stable, well-tolerated dose for the previous 3 months with no further changes anticipated
* Agrees not to discuss treatment outcomes on social media until subject has completed their End of Therapy visit

Exclusion Criteria:

* Active or history of peptic or gastric ulcer or hemorrhage
* Any chronic major medical comorbid condition deemed by the Investigator as presenting added risk to the subject, including but not limited to refractory hypertension, kidney disease, or liver disease
* Diagnosed with diabetes (Type 1 or II) or receiving any anti-diabetic medication
* Unstable seizure disorder defined by any seizure within 6 months prior to baseline visit and/or a change in any anti-convulsant drug dosing in the 60 days prior to study entry
* Patients with cardiovascular disease risk factors: Uncontrolled high blood pressure (systolic blood pressure >150 mmHg), Unstable angina, History of documented myocardial infarction or cerebrovascular accident, NYHA Class III and IV heart failure, Known uncontrolled hyperlipidemia as LDL-C ≥190 mg/dL or triglycerides ≥ 500 mg/dL
* Chronic use of NSAIDs or other anti-inflammatory agents
* Currently taking or have taken any cannabidiol (CBD) preparation within 30 days prior to screening
* Currently taking or have taken sulindac or gaboxadol within 30 days prior to screening
* Currently taking GABAergic agents (i.e., acamprosate, baclofen, vigabatrin, tiagabine, riluzole, benzodiazepines, and gabapentin)
* Changes in psychotropic or anti-convulsant (where taken for reasons other than seizure control) drug treatment within 30 days prior to Screening
* Significant changes in any educational, behavioral and/or dietary interventions the month prior to Screening
* Planned initiation of new, or modification of ongoing, interventions during the study
* History of adverse effects of sulindac or other NSAIDs that would prevent safe study completion
* Unable or unwilling to take oral medication (whole capsule) or history of dysphagia or malabsorption
* Has abnormal baseline laboratory assessments including, but not limited to, ALT or AST or total bilirubin >1.5 × ULN, or other clinically relevant laboratory abnormality
* Has a clinically significant abnormal ECG, heart rate or BP at Screening as judged by the Investigator
* Has received an investigational drug (either approved or not approved) in any prior clinical study within 30 days or 5 half-lives (whichever is longer) prior to Screening

Ages: 13 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
NIH Cognitive Toolbox | Day 70
Clinical Global Impression - I | Day 70
Aberrant Behavior Checklist | Day 70
Anxiety, Depression, and Mood Scale | Day 70
FXS Domain Specific Concerns | Day 70
  The Clinician/Caregiver FXS Domain Specific Concerns allows for the subject specific symptoms of concern to be assessed on an ongoing basis throughout the study. The specific concerns that correlate to the 6 domains (Clinician) or 3 Domains (Caregiver) will be assessed using a 7-point Likert scale.

SECONDARY OUTCOMES:
To assess the safety and tolerability of each dose | Day 70
  Incidence of adverse events (AEs) and serious adverse events (SAEs) reported during the study. Change from baseline to Day 70 in physical examinations and assessment of vital signs.
Kiddie Test of Attentional Performance (KiTAP) | Day 70
Emotional Faces Tobii Eye Tracking | Day 70
EEG | Day 70
  Resting state whole brain EEG spectra activity in 3 EEG assessments (EEG spectra, auditory evoked response potential (ERP) and Chirp modulated sweep.
CGI-S | Day 70

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Berry-Kravis, Principal Investigator — Rush University Medical Center & Children's Hospital
Locations (10):
- United States (7):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Rush University Medical Center & Children's Hospital, Chicago, Illinois
  - Kennedy Krieger Insitute, Baltimore, Maryland
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Icahn School of Medicine (Mount Sinai), New York, New York
- Australia (3):
  - Children's Health Queensland Hospital and Health Service, Brisbane, Queensland
  - Fragile X Alliance Clinic, Caulfield, Victoria
  - Murdoch Children's Research Institute, Melbourne, Victoria